CLINICAL TRIAL: NCT02768623
Title: Evaluation of a Community Pharmacist Managed Asthma Consultation Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zahava Rosenberg-Yunger (Other)
Responsible Party: Sponsor-Investigator, Zahava Rosenberg-Yunger, Dr. Rosenberg-Yunger, Toronto Metropolitan University
Organization: Toronto Metropolitan University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RyersonU1
Record Dates: First submitted 2016-03-08; First posted 2016-05-11 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Uncontrolled Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Active Comparator): Patients in the control group will receive standard, dispensing services they currently receive from pharmacists. Control group pharmacists will continue to provide these services in accordance with the standards of practice adopted by the Ontario College of Pharmacists. They will not provide either of the 3 intervention components outlined above. Should a control group patient request additional information and/or services, the pharmacist will comply and provide these as deemed necessary for the particular patient. This could include the full range of educational and drug therapy optimization services outlined for the intervention group. If this occurs then the pharmacists will document all services provided in order for the research team to account for this in the analysis.
  Interventions: Other: Pharmacist Intervention (when requested by patient)
- Intervention Group (Experimental): Pharmacists in the intervention group will provide patients with a comprehensive disease management program for asthma. The 3 major components of pharmacists' intervention are outlined below. The services delivered will be customized based on each patient's case.
  1. Medication review and drug therapy optimization
  2. Patient education
  3. Improving patient adherence
  Interventions: Other: Pharmacist led Asthma Management

INTERVENTIONS:
Other: Pharmacist led Asthma Management
  Other Names: Pharmacist Asthma Intervention
  Arms: Intervention Group
Other: Pharmacist Intervention (when requested by patient)
  Arms: Control Group

SUMMARY:
Asthma is one of the most common chronic health conditions, affecting 900,000 Ontarians, 2.4 million Canadians and over 300 million people worldwide. Unlike most other chronic diseases, asthma affects a significant proportion of children - an estimated 21% in Ontario. Asthma is also the leading cause of hospitalization for children in Canada and is a significant cause of school and work absenteeism. Though asthma is generally considered a chronic disease, it can be fatal in some instances - in 2009, an estimated 91 Ontarians died of this condition. Effective management of asthma can prevent exacerbation and more severe negative health consequences. In fact, estimates show that over 80% of the asthma-related deaths could be prevented through proper education. However, evidence also shows that over 55% of patients with moderate to severe asthma do not have their asthma symptoms under control, despite regular doctor visits. Less than a third (31%) of asthma patients report receiving an asthma action plan from their physicians, although such plans are associated with fewer ER visits, lower hospitalization rates and improved lung function. Hence, there is a clear opportunity to improve the management of asthma and reduce the incidence of related complications.

Given the scientific evidence of pharmacists effect on asthma management there is a strong rationale for introducing an asthma-specific pharmacist-led intervention for Ontarians suffering from this chronic disease. However, the implementation of such a program should be preceded by a pilot test to ensure that the program parameters are optimized to drive improved patient outcomes and maximum quality of service. The primary goals of this research project are to examine the impact of a pharmacist led asthma management intervention on patient health outcomes and to determine the optimum program structure to ensure quality of service delivery.

This study employs a mixed-methods study design. Investigators will begin with a cluster randomized controlled trial and end with exit interviews.This study will consist of a prospective, randomized controlled trial conducted in the community setting. A total of 12 pharmacies across the Greater Toronto Region will be recruited for this study. Each of these pharmacies will be randomly assigned in a 1:1 ratio to either the intervention group or the control group. All data will be analyzed using statistical software. Significance level will be set at 0.05. Pharmacy level descriptive characteristics, including mean and standard deviation for the number of patients will be reported. There is a low perceived risk for this study; however, the investigators will take every precaution to ensure this study is conducted in an ethical manner, including protecting patient confidentiality and anonymity.

ELIGIBILITY:
Inclusion Criteria:

* Provided written consent
* Intending to refill all asthma-related prescriptions at the study pharmacy
* Diagnosed with asthma by a physician or nurse practitioner
* Taking inhaled corticosteroids for which the dose and/or medication has remained unchanged for at least 2 months
* 18 years of age or older
* Uncontrolled asthma (defined as in the past 4 weeks the patient has used their rescue medications 4 or more times in a given week and/or the patient has woken up in the night from their asthma in a given week).

Exclusion Criteria:

* Pregnant women
* Unable or unwilling to return to the pharmacy for scheduled visits
* Unable to speak English language well enough to communicate with the pharmacist and complete the questionnaires independently
* Terminal illness or poor prognosis (life expectancy less than 3 years)
* History of alcoholism or drug abuse
* Comorbidities/health issues:

  * Chronic obstructive pulmonary disorder (emphysema; chronic bronchitis)
  * Acute respiratory infection
  * Pulmonary fibrosis
  * Cancer (in the past 5 years preceding enrolment)
  * Organ transplantation
  * Dementia, cognitive impairment or other psychiatric disorder (Cognitive Impairments such as those found under the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) common Axis I and Axis II disorders
  * Any other health issue that may hinder performance on pulmonary function test
* Enrolled in an Employee Assistance Program for disease management within 6 months preceding the study enrolment date OR planning to enroll in the next 12 months
* Enrolled in another asthma management/clinical study OR planning to enroll in a similar study in the next 12 months
* Had a MedsCheck or MedsCheck Follow-Up done within the 3-month period preceding the anticipated date of the first study appointment
* Patients who do not wish their physician to be notified of their participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
Peak Expiratory Flow Rate (PEF) | Pharmacist will measure peak flow rate incrementally each month for 12 months total.
  A peak flow meter will be used to measure PEF.

SECONDARY OUTCOMES:
Peak Flow Diary | Patients will measure their peak flow twice daily (morning and night) throughout the duration of the study (i.e., 12 months) with their peak flow meter. They will document their peak flow measurements in a diary.
  The peak flow diary is a chart given to patients to assist in recording their peak flow measurement using the peak flow meter.
Asthma Control | Pharmacist will measure Asthma control twice throughout duration of study. First, it will be measured at baseline (month 1) and lastly it will be measured at the final appointment (12 months after baseline).
  The Asthma Control Questionnaire will be used to measure Asthma Control.
The Medication Adherence Report Scale for Asthma | Pharmacist will measure Medication Adherence twice throughout duration of study. First, it will be measured at baseline (month 1) and lastly it will be measured at the final appointment (12 months after baseline).
  The Medication Adherence Report Scale for Asthma will be used to measure adherence to asthma medication.
Health Care Service Usage Questionnaire | Pharmacist will measure Health Care Service Usage twice throughout duration of study. First, it will be measured at baseline (month 1) and lastly it will be measured at the final appointment (12 months after baseline).
  The Health Care Service Usage Questionnaire will be used to measure a patient's utilization of health care services.
Asthma Quality of Life Questionnaire (AQLQ) | Pharmacist will measure Asthma related quality of life twice throughout duration of study. First, it will be measured at baseline (month 1) and lastly it will be measured at the final appointment (12 months after baseline).
  The AQLQ will be used to measure patient's quality of life.
Heath and Work Performance Questionnaire | Pharmacist will measure health and work performance twice throughout duration of study. First, it will be measured at baseline (month 1) and lastly it will be measured at the final appointment (12 months after baseline).
  The Heath and Work Performance Questionnaire will be used to measure patient's presenteeism and absenteeism due to asthma.
Asthma Self-Management Questionnaire | Pharmacist will measure Asthma self-management twice throughout duration of study. First, it will be measured at baseline (month 1) and lastly it will be measured at the final appointment (12 months after baseline).
  The Asthma Self-Management Questionnaire will be used to assess the patient's asthma management techniques.
Asthma General Knowledge Questionnaire for Adults | Pharmacist will measure Asthma general knowledge twice throughout duration of study. First, it will be measured at baseline (month 1) and lastly it will be measured at the final appointment (12 months after baseline).
  The Asthma General Knowledge Questionnaire for Adult will be used to assess patient's asthma knowledge.
Patient Satisfaction Questionnaire | The pharmacist will distribute this questionnaire to patients at the final appointment (12 months after baseline).
  The Patient Satisfaction Questionnaire will be used to assess patients' satisfaction with the services they received over the study duration.

CONTACTS AND LOCATIONS:
Overall Officials: Zahava Rosenberg-Yunger, PhD, Principal Investigator — Ryerson University; Ontario Pharmacists Association